CLINICAL TRIAL: NCT00054353
Title: Reduced-Intensity Allogeneic HSC Transplantation From HLA-Matched Related and Unrelated Donors for Patients With Multiple Myeloma - A Multi-Center Trial
Brief Title: Reduced-Intensity Conditioning Followed By Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marco Mielcarek, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1743.00; NCI-2011-00386 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1743.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine phosphate; Melphalan; Whole-Body Irradiation; Mycophenolic Acid; Cyclosporine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Related Donor (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -3 and intermediate-dose melphalan IV over 15-20 minutes on day -2. Patients also undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 80 with taper to day 180 (related donors) or on days -3 to 100 with taper to day 180 (unrelated donors). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related donors) or TID on days 0-40 with taper to day 96 (unrelated donors).
  Interventions: Drug: fludarabine phosphate; Drug: melphalan; Radiation: total-body irradiation; Drug: mycophenolate mofetil; Drug: cyclosporine; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis
- Unrelated Donor (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -3 and intermediate-dose melphalan IV over 15-20 minutes on day -2. Patients also undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 80 with taper to day 180 (related donors) or on days -3 to 100 with taper to day 180 (unrelated donors). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related donors) or TID on days 0-40 with taper to day 96 (unrelated donors).
  Interventions: Drug: fludarabine phosphate; Drug: melphalan; Radiation: total-body irradiation; Drug: mycophenolate mofetil; Drug: cyclosporine; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo reduced-intensity allogeneic PBSCT
Procedure: peripheral blood stem cell transplantation — Undergo reduced-intensity allogeneic PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects of giving reduced-intensity conditioning followed by donor peripheral blood stem cell transplant (PBSCT) and how well it works in treating patients with multiple myeloma (MM). Giving low doses of chemotherapy, such as fludarabine phosphate and melphalan, and total-body irradiation (TBI) before a donor PBSCT helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving mycophenolate mofetil and cyclosporine after transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of this approach by determining the 1-year progression-free survival (PFS) and overall survival (OS).

II. To evaluate day 100 non-relapse mortality.

III. To determine the incidences of grades II-IV acute graft-versus-host disease (GVHD) and chronic extensive GVHD.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -5 to -3 and intermediate-dose melphalan IV over 15-20 minutes on day -2. Patients also undergo low-dose TBI on day 0.

TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) on days -3 to 80 with taper to day 180 (related donors) or on days -3 to 100 with taper to day 180 (unrelated donors). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related donors) or thrice daily (TID) on days 0-40 with taper to day 96 (unrelated donors).

After completion of study treatment, patients are followed up at 3, 6, 12, 18, and 24 months, and then annually thereafter for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Meet Salmon and Durie criteria for initial diagnosis of MM; transplant will be offered to patients with previously treated MM who meet one of the following criteria:

  * Patient received at least one prior autologous or syngeneic hematopoietic SCT (HSCT) and now has progressive disease (PD) (greater than 25% increase in serum or urine paraprotein levels compared to best response status after autograft or appearance of new lytic bone lesions or plasmocytomas)
  * Patient is not able to collect autologous PBSC due to poor marrow reserve (insufficient HSC-mobilization: < 2.5 x 10^6 cluster of differentiation [CD]34+ cells/kg); or contraindications to undergoing HSC-mobilization; patient now has PD and has received at least 4 cycles of standard chemotherapy (e.g. vincristine sulfate, doxorubicin hydrochloride, and dexamethasone [VAD]) in the past
* Patients must have the capacity to give informed consent
* DONOR: Human leukocyte antigen (HLA) genotypically identical sibling or phenotypically matched relative
* DONOR: HLA phenotypically matched unrelated donor (according to Standard Practice HLA matching criteria)

  * Matched for serologically recognized HLA-A or B or C antigens and at least five of six HLA-A or B or C alleles
  * Matched for HLA DRB1 and DQB1 alleles (defined by high-resolution typing) at the allele level
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis for PBSC collection
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of a temporary central venous catheter

Exclusion Criteria:

* Karnofsky score < 60%
* Left ventricular ejection fraction < 40% or symptomatic heart failure; ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL,or symptomatic biliary disease
* Diffusion capacity of carbon monoxide (DLCO) < 50% (corrected) or receiving continuous supplemental oxygen
* Creatinine clearance < 40 mL/min
* Patients with poorly controlled hypertension
* Seropositive for the human immunodeficiency virus (HIV)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Pregnancy or breastfeeding
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Not fully recovered from previous high-dose therapy:

  * Persistent mucositis and gastrointestinal symptoms requiring hyperalimentation and/or intravenous hydration
  * On steroids for autologous/syngeneic GVHD
  * On IV antibiotics for documented infections
  * Cytomegalovirus (CMV)-antigenemia positive
  * On ganciclovir or foscarnet for previous CMV reactivation/infection; off of this therapy for less than two weeks despite documented CMV-antigenemia- negativity (identification [ID] should be consulted if there is persistent CMV antigenemia post autograft)
  * Ongoing radiotherapy
  * Patients who meet any of these criteria may be discussed with the principal investigator for recommendations as to the timing of the allograft
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* DONOR: Identical twin
* DONOR: Donors unwilling to donate PBSC
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness
* DONOR: Failure to meet Fred Hutchinson Cancer Research Center (FHCRC) criteria for stem cell donation
* DONOR: Age < 12 years
* DONOR: A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-10; Primary Completion 2009-10 (Actual); Study Completion 2012-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mielcarek, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States
- University of Torino, Torino, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Related Donor; Unrelated Donor: PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -3 and intermediate-dose melphalan IV over 15-20 minutes on day -2. Patients also undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 80 with taper to day 180 (related donors) or on days -3 to 100 with taper to day 180 (unrelated donors). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related donors) or TID on days 0-40 with taper to day 96 (unrelated donors).
  fludarabine phosphate: Given IV melphalan: Given IV total-body irradiation: Undergo TBI mycophenolate mofetil: Given PO
  cyclosporine: Given PO
  nonmyeloablative allogeneic hematopoietic stem cell transplantation: Undergo reduced-intensity allogeneic PBSCT
  peripheral blood stem cell transplantation: Undergo reduced-intensity allogeneic PBSCT
  laboratory biomarker analysis: Correlative s
Period: Overall Study
Arm/Group | Related Donor | Unrelated Donor
Started | 12 | 4
Completed | 12 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Related Donor | Unrelated Donor | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 3 | 13
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 4 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12
  Italy | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: PFS will be calculated for all patients from the date of transplant until the time of progression, relapse, death, or the date the patient was last known to be in remission. Progressive disease is defined as greater than 25% increase in serum or urine M proteins compared to best response status after autologous transplant and/or appearance of new lytic bone lesions or plasmocytomas.
Time Frame: At 1 year post-transplant
Population: There were 4 patients who, although they did not have progression/relapse, died before the 1 year mark, and thus are not included in the 1 year PFS count.
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 9 | 3
Participants | 4 | 1

2. Primary Outcome: Non-relapse Mortality
Description: Early NRM will be monitored in a sequential fashion.
Time Frame: At day 100
Measure: Count of Participants; unit: Participants
Groups:
- Related Donor; Unrelated Donor: PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -3 and intermediate-dose melphalan IV over 15-20 minutes on day -2. Patients also undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 80 with taper to day 180 (related donors) or on days -3 to 100 with taper to day 180 (unrelated donors). Patients also receive mycophenolate mofetil PO BID on days 0-27 (related donors) or TID on days 0-40 with taper to day 96 (unrelated donors).
  fludarabine phosphate: Given IV melphalan: Given IV total-body irradiation: Undergo TBI mycophenolate mofetil: Given PO cyclosporine: Given PO
  nonmyeloablative allogeneic hematopoietic stem cell transplantation: Undergo reduced-intensity allogeneic PBSCT
  peripheral blood stem cell transplantation: Undergo reduced-intensity allogeneic PBSCT
  laboratory biomarker analysis: Correlative studies
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants | 1 | 1

3. Primary Outcome: Incidence of Acute GVHD (Grades III-IV)
Description: Number of patients with Grade III-IV acute GVHD post-transplant. Severe GVHD will be monitored in a sequential fashion.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants | 2 | 0

4. Primary Outcome: Incidence of Chronic (Extensive) GVHD
Description: Number of subjects with chronic extensive GVHD post-transplant. Severe GVHD will be monitored in a sequential fashion.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants | 4 | 1

5. Secondary Outcome: OS
Description: Number of subjects surviving. OS will be estimated by the method of Kaplan and Meier. Confidence intervals will be estimated.
Time Frame: At 6 months and then every year thereafter, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants
  6 Months | 8 | 3
  1 Year | 5 | 2
  2 Years | 4 | 0
  3 Years | 3 | 0
  4 Years | 3 | 0
  5 Years | 3 | 0

6. Secondary Outcome: Engraftment
Description: Number of subjects who engrafted post-transplant. Engraftment will be monitored in a sequential fashion.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants | 12 | 4

7. Secondary Outcome: Relapse Rate
Description: Number of subjects who relapsed after achieving CR post-transplant. Relapse rate will be summarized using cumulative incidence estimates.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants | 1 | 1

8. Secondary Outcome: Response Rate
Description: Number of subjects who achieved CR post-transplant. Response rate will be summarized using cumulative incidence estimates.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donor | Unrelated Donor
Number analyzed (Participants) | 12 | 4
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Related Donor | Unrelated Donor
All-Cause Mortality (participants affected / at risk) | 4/12 | 1/4
Serious Adverse Events (participants affected / at risk) | 4/12 | 1/4
Other Adverse Events (participants affected / at risk) | 9/12 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Related Donor (N=12) | Unrelated Donor (N=4)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Related Donor (N=12) | Unrelated Donor (N=4)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Generalized muscle weaknes (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes